CLINICAL TRIAL: NCT00982059
Title: Colorectal Cancer Screening in Cancer Survivors Treated With Radiation Therapy
Brief Title: Colorectal Cancer Screening for Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 07-0708-CE
Record Dates: First submitted 2008-11-21; First posted 2009-09-22 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; Cancer survivor; Radiation therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All: All patients enrolled in the study will be undergoing the same procedures.
  Interventions: Other: Colonoscopic examination

INTERVENTIONS:
Other: Colonoscopic examination — All patients enrolled in the study will undergo a colonoscopic examination and complete a baseline questionnaire.

SUMMARY:
The risk of colorectal cancer (CRC) is significant among cancer survivors treated with abdominal radiation therapy (RT). Further, CRC is once of the few cancers for which there is effective screening. Although some expert groups recommend early CRC screening for patients with prior abdominal RT, the effectiveness of early screening is unknown. It is also unknown if radiation-induced CRC passes through a "pre-clinical" phase in which precancerous polyps are detectable and treatable prior to becoming invasive cancers. This study will evaluate whether screening will detect pre-invasive colorectal polyps among survivors treated with RT.

DETAILED DESCRIPTION:
Cancer survivors meeting the COG criteria for CRC screening will undergo colonoscopy and removal of colorectal polyps. Documentation of polyp number, location and pathologic characteristics will be made. Clinical data information will also be collected at the time of patient enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic survivors treated with ≥ 25Gy to the abdomen, pelvis or spine, or ≥ 12Gy total body radiation therapy, or ≥ 12Gy whole abdominal RT.
2. Patients who have passed ≥10 years following RT
3. Patients whose current age is 35-49.

Exclusion Criteria:

1. Patients with signs/symptoms suggestive of CRC or other high-risk features such as:

   * Persistent constipation for >2 weeks in the last month
   * One or more unexplained episodes of red blood in the stool in the last month
   * One or more unexplained episodes of black stool in the last month
   * Unexplained pelvic pain in the last month
2. Patients with a history of Crohn's disease or ulcerative colitis
3. Patients already taking part in a colorectal screening program defined as any colorectal screening (colonoscopy, sigmoidoscopy, fecal occult blood test) within last 5 years.
4. Patients with self-reported history of colorectal polyps.

Ages: 35 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have received radiation treatment to the abdomen,pelvis or spine.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2008-05; Primary Completion 2014-12 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
The proportion of screened patients with any polyp or any high risk polyp will be calculated. | 3 years

SECONDARY OUTCOMES:
Proportion calculation/identification of: demographic/treatment influences on polyp prevalence; subgroups w/polyp prevalence >20%; pts with polyps beyond 30cm flexible sigmoidoscope; pts with adenomatous polyp(s) on colonoscopy in/outside prior RT fields | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Hodgson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital; Andrea K Ng, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Daly PE, Samiee S, Cino M, Gryfe R, Pollett A, Ng A, Constine LS, Hodgson DC. High prevalence of adenomatous colorectal polyps in young cancer survivors treated with abdominal radiation therapy: results of a prospective trial. Gut. 2017 Oct;66(10):1797-1801. doi: 10.1136/gutjnl-2016-311501. Epub 2016 Jul 13. PMID 27411369